CLINICAL TRIAL: NCT06239285
Title: A Virtual Reality Brief Violence Intervention: Preventing Gun Violence Among Violently Injured Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20027823_Thomson; R01CE003625 (NIH)
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Violence
Keywords: Firearm Violence Victim
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A randomized control trial (RCT) in a large sample of violently injured adults (18+ years) from VCU Health.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) Group (Placebo Comparator): The treatment-as-usual (TAU) group will receive a community resource brochure (the same one that is provided at the end of BVI-VR). This brochure provides contact detail for services in the local area.
  Interventions: Other: Treatment as Usual (TAU)
- Intervention Group (Experimental): Patients randomized into the BVI-VR group will answer questions about the session content and the rationale for the content. Their responses will provide an estimate of engagement providing a better understanding of treatment fidelity.
  Interventions: Device: Brief Violence Intervention VR (BVI-VR)

INTERVENTIONS:
Device: Brief Violence Intervention VR (BVI-VR) — BVI-VR is being developed as a hospital-based brief gun violence intervention program founded on the principles of positive psychology, motivational goal setting (via gameplay), psychoeducation, cognitive-behavioral therapy, and dialectical behavioral therapy. All steps of the BVI-VR emphasize being in control of making positive choices, and how to locate and leverage opportunities within their communities to improve their well-being. BVI-VR empowers patients to be the driver of their well-being
  Arms: Intervention Group
Other: Treatment as Usual (TAU) — group will receive a community resource brochure (the same one that is provided at the end of BVI-VR). This brochure provides contact detail for services in the local area. These include organizations that provide mental health counseling, mentorship services, career development programs, organized community activities and sports, educational support, financial support, substance abuse programs, and resource assistance (e.g., food, housing, etc.).
  Arms: Treatment as Usual (TAU) Group

SUMMARY:
The overall aim of the proposed project is to develop and evaluate the effectiveness of Brief Violence Intervention-Virtual Reality (BVI-VR) for reducing firearm-related violence, re-injury, and mortality among victims of violence. Outcome measures of firearm-related violence will come from multiple sources, including criminal background checks, hospital data, state-level data, semi-structured clinical assessments, and self-report assessments. In addition, the study aims to understand the impact of BVI-VR on psychosocial mediators resulting in a reduction of firearm-related violence. This will include self-report surveys, neurocognitive assessments, and clinical assessments. The economic efficiency of BVI-VR as a firearm-related violence intervention will also evaluated. To achieve these aims, a randomized control trial (RCT) in a large sample of violently injured adults (18+ years) from VCU Health will be conducted.

DETAILED DESCRIPTION:
Brief Violence Intervention-Virtual Reality (BVI-VR) is being developed as a hospital-based brief gun violence intervention program founded on the principles of positive psychology, motivational goal setting (via gameplay), psychoeducation, cognitive-behavioral therapy, and dialectical behavioral therapy. This proposal will develop five steps to create a 30-minute brief firearm-related violence intervention. The five steps address a range of psychosocial risk factors and enhance protective factors for violence, as well as psychoeducational programming specifically addressing the risk of firearm violence. All steps of the BVI-VR emphasize being in control of making positive choices, and how to locate and leverage opportunities within their communities to improve their well-being. BVI-VR empowers patients to be the driver of their well-being.

ELIGIBILITY:
Inclusion Criteria:

* violently injured patients from VCU's Level 1 Trauma Center
* 18 years or older
* English-speaking

Exclusion Criteria:

* Under 18 years old
* Not a victim of Violent crime

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Firearm-related violence /The gun violence questionnaire | Baseline self-report, 3- and 6-months post-randomization
  The gun violence questionnaire is a 9-item self-report that assesses firearm-related violence. Items were adapted from the Buss-Perry Aggression Questionnaire physical aggression scale; for example, "Given enough provocation, I may fire my gun at another person". The measure has adequate internal consistency (α = .75) and good convergent and discriminant validity with other violence related measures
Gun Behaviors and Beliefs Scale | 3 and 6 month post baseline
  Gun Behaviors and Beliefs Scale will be used to measure gun behaviors and beliefs that may be impacted by the intervention: Safety and Control, Social Perceptions, Emotional Risk, Common Beliefs. The subscales have demonstrated adequate to good internal consistency (α = .79-.96).
Firearm criminal conviction and arrests/ Criminal Background Checks | prior to baseline assessment, from baseline to 3-month follow-up, and from 3-month follow-up to the 6-month follow-up.
  Criminal background checks will be conducted on participants to assess violent criminal arrests and gun-related crimes and police contacts. Criminal activity will be coded for the occurrence of nonviolent crime, violent crime, and firearm-related crime for three-time points: prior to baseline assessment, from baseline to 3-month follow-up, and from 3-month follow-up to the 6-month follow-up.
Non-convicted firearm-related violent crime/ Violent Crime Assessment | 3 and 6 month post baseline
  Violent Crime Assessment is a semi-structured clinical assessment of convicted and non-convicted violent crime. The measure captures six categories of violent crimes that participants have and have not been arrested for; simple assault, aggravated assault, homicide, robbery, rape, and sexual assault. Information is collected on weapon use for each of the crimes (e.g., used a firearm during rape; fired a gun at a party and may have hit someone). The VCA provides a valuable index for firearm-related violence that is not captured in self-report measures or criminal background checks.

SECONDARY OUTCOMES:
Firearm-related re-injury/ Self-report | 3 and 6 month post baseline
  Violent injury data are collected from self-report surveys which capture the number of times a participant has been violently injured and what the patient was injured by (GSW).
Firearm-related re-injury/ Hospital data: Virginia Department of Health | 3 and 6 month post baseline
  Violent injury data are collected from VCU's hospital database.
Firearm-related mortality/ Hospital data; Virginia Department of Health; National Death Index | 3 and 6 month post baseline
  Mortality rates will be collected from hospital records and the National Death Index database.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Thomson, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided